CLINICAL TRIAL: NCT03816722
Title: The Effect of High Flow, Nasal Cannula Delivered Air in Patients With Interstitial Lung Disease - a Pilot Study
Brief Title: High Flow in Interstitial Lung Disease
Acronym: HiFloILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Ulla Møller Weinreich, Principal Investgator, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: N-20180070
Record Dates: First submitted 2018-12-06; First posted 2019-01-25 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Prospective, unblinded cross over study
Masking Description: As blinding of high flow treatment in not possible this is an open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): Patients starting the cross over with 6 weeks of high flow treatment with Airvo2 in addition to usual care
  Interventions: Device: Airvo2; Other: Usual care
- control (Experimental): Patients starting the cross over in the usual care Group but after 6 weeks receiving High Flow treatment with Airvo2
  Interventions: Device: Airvo2; Other: Usual care

INTERVENTIONS:
Device: Airvo2 — Treatment with HighFlow through the Airvo2 device, 8 hours per day
Other: Usual care — High flow treatment is investigated as an add on treatment to the personalized care already prescribed to the patients. As patients with interstitial lung disease very often demand very different treatment set ups treatment will vary in the individual patients. All will, however, be treated with ambulatory oxygen. "Usual care" will be unaltered a month before inclusion in the study in each of the individual patients
  Other Names: Ambulatory oxygen therapy, personalised medicine

SUMMARY:
This is a prospective, 6 week cross-over study on the effect of High flow nasal cannula (HFNC) delivered air in patients with interstitial lung disease (ILD), in need of ambulatory oxygen therapy.

Primary outcome:

To investigate intra-personal differences in 6MWT, as well as SO2 and BORG score at the end of the 6MWT, at baseline, at 6 weeks and 12 weeks To investigate intra-personal differences in SGRQ at baseline, at 6 weeks and 12 weeks To investigate intra-personal differences in quality of sleep, using the Richards-Campbell sleep questionnaire (RCSQ) at baseline, at 6 weeks and 12 weeks To investigate intra-personal differences in IC, at baseline, at 6 weeks and 12 weeks

Secondary outcome:

To investigate intra-personal differences in FVC, at baseline, at 6 weeks and 12 weeks To investigate intra-personal differences in DLCO at baseline, at 6 weeks and 12 weeks To investigate intra-personal differences in mMRC-score at baseline, at 6 weeks and 12 weeks

DETAILED DESCRIPTION:
In this pilot study we wish to investigate whether treatment with HFNC, delivered by MyAirvo2 (Fisher&Paykel, Auckland, New Zealand) in patients with interstitial lung disease (ILD) in need of ambulatory oxygen therapy (AOT).

Ten patients will be recruited from the outpatient clinic at Department of Respiratory Diseases, Aalborg University Hospital.

The study is carried out as a cross over study, randomizing 5 patients to intitially 6 weeks' HFNC treatment as add on to the patients' personalized usual care followed by 6 weeks observation on usual care and 5 patients to 6 weeks' observation on the patients' personalized usual care, followed by 6 weeks with HFNC as add on to usual care.

At inclusion patients' background information will be registered and patients will be examined with body plethysmography, registering TLC, FVC, RV and IC, as well as DLCO. Furthermore, a 6MWT will be performed, monitoring peripheral oxygen saturation (SO2)and BORG score at the beginning and the end of the procedure as well as analysis of arterial blood gasses (PaO2, PaCO2) at rest. In addition the modified Medical Research Council (mMRC)- score; the Richards-Campbell Sleep Questionaire (RCSQ) and the St. George Respiratory Questionaire (SGRQ) will be carried out at baseline. Following this, patients will be randomized to either usual care or usual care plus HFNC, recommended flow 30 liters/minute, recommended temperature 37o Celsius, recommended use 8 hours/day, preferably at night. After 6 weeks body plethysmography, 6MWT, mMRC, SGRQ, RCSQ and arterial blood gas analysis will be repeated and following this, treatment will cross over; as such, patients initially in the usual care arm will be treated with HFNC as add on according to the recommendations stated above and the previous HFNC treated group will be referred to usual care for the following 6 weeks. At the end of the study period (t=12 weeks), body plethysmography, 6MWT, mMRC, RCSQ, SGRQ and arterial puncture will be repeated in all patients as well as background information will be revisited to note any changes.

Should the patient reach chronic respiratory failure (saturation at rest < 88%) during the study period, patients will remain in study and the airflow during HFNC be oxygenated with whatever amount of oxygen is required to reach saturation >88% during High Flow treatment.

Equipment:

Heated, humidified, air will be delivered to the patients by MyAirvo 2 (Fisher&Paykel, Auckland, New Zealand). Patients will be treated with an intended flow of 30 L/min, intended use 8 hours per day, preferably nocturnal use. Should patients not tolerate the recommended flow, changes in flow are allowed. The Airvo2 device will be delivered and serviced in the patients' homes by VitalAire. Vitalaire will do readings of actual use on the device. At the end of the study, all patients will be offered continuous treatment with the device if so desired.

ELIGIBILITY:
Inclusion criteria

* Age > 18 years old
* Patient diagnosed with interstitial lung disease
* Capable of understanding oral and written information and giving informed consent
* Newly diagnosed with need of oxygen during physical activity (SO2 <88%).

Exclusion criteria

* Pneumonia or exacerbation of ILD < 6 weeks prior to inclusion
* Other terminal disease than ILD and life expectancy < 3 months
* Patients not capable of understanding and accepting written or verbal information
* Patients with in need of continuous oxygen treatment at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | change between 6 and 12 weeks
  walking distance
SO2 | change between 6 and 12 weeks
  oxygen saturation of the blood
modified BORG score | 6 and 12 weeks
  score of dyspnea, ranging 0-10 where 0 is no dyspnea
St George Respiratory Questionaire (SGRQ) | change between 6 and 12 weeks
  respiratory quality of life questionnaire, score with 20 questions all weighted in the final evaluation of the score. A change of 4 points is clinically relevant; a change of -4 an amelioration of quality of life
Richards-Campbell's sleep questionnaire (RCSQ) | change between 6 and 12 weeks
  Quality of sleep questionnaire, based on 5 domains, evaluated individually by Visual Analog Scores(0-100), where 0 is the worst, 100 is the best outcome. All scores are equally weighted in the final score. The final, combined score is averaged, and expressed as a percentage of the total score
inspiratory capacity | change between 6 and 12 weeks
  lung function measure (L, %)

SECONDARY OUTCOMES:
Forced Vital Capacity | change between 6 and 12 weeks
  lung function measure (L, %)
diffusion capacity of the lung for carbon monoxide (DLCO) | change between 6 and 12 weeks
  diffusion capacity measure, (% of expected value)
modified Medical Research Council score (mMRC-score) | change between 6 and 12 weeks
  dyspnea-score, scoring from 0-4 points

CONTACTS AND LOCATIONS:
Overall Officials: Ulla M Weinreich, MD, PhD, Principal Investigator — Aalborg University Hospital, Mølleparkvej 4, 9100 Aalborg, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
There a no IPD sharing plans at present